CLINICAL TRIAL: NCT01364909
Title: Early Intervention With Exercise in Critically Ill Patients With Sepsis: a Randomized Controlled Trial
Brief Title: Exercise in Critically Ill Patients With Sepsis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Queensland (Other)
Collaborators: Royal Brisbane and Women's Hospital (Other Government)
Responsible Party: Dr Jennifer Paratz, The University of Queensland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XSEP1
Record Dates: First submitted 2011-05-27; First posted 2011-06-03 (Estimated); Last update posted 2011-06-03 (Estimated); Status verified 2008-10

CONDITIONS: Sepsis Syndromes
Keywords: Sepsis; Severe sepsis; Septic shock; Septicaemia; Bacteremia
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Sepsis; Shock, Septic; Toxemia; Bacteremia | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (usual practice) (Placebo Comparator)
  Interventions: Other: Usual practice
- Exercise (Experimental)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — The subjects will be given 2 x 30 minute sessions of exercise per day consisting of either passive, active, active assisted depending on level of sedation and stability of condition.
  According to level of sedation and stability they may also perform sitting exercises
  Arms: Exercise
Other: Usual practice — These patients will not receive exercise early in their intensive care admission
  Arms: Control (usual practice)

SUMMARY:
This study will investigate whether early exercise in critically ill patients will decrease inflammatory markers, increase pro-inflammatory markers and prevent loss of muscle mass.

DETAILED DESCRIPTION:
This study will investigate the effects of an early targeted rehabilitation program on inflammatory markers and muscle mass in patients with sepsis syndromes in intensive care.

The Primary Hypothesis is that an early targeted rehabilitation ICU patients with sepsis syndromes over 7 days will Prevent loss of lean muscle mass by within 7 days of recruitment to the study. Decrease pro-inflammatory and increase anti-inflammatory cytokines within 7 days of recruitment to the study.

ELIGIBILITY:
Inclusion Criteria:

* Systemic inflammatory response syndrome with a proven or suspected infectious etiology.
* 18 years and over
* Relatives willing to give consent
* Admitted to intensive care and likely to remain ventilated for > 48 hours

Exclusion Criteria:

* Patients with septic shock unresponsive to maximal treatment or who are moribund or have an expected mortality within 48 hours
* Head injuries
* Burn injury
* Multiple lower limb fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-06; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Fat free mass ie muscle mass (lean tissue) | Change from baseline to one week, then change from baseline to two weeks
  Fat free mass will be measured by Multi-Frequency Bioelectrical Impedance Spectroscopy (BIS) (ImpediMed SFB7, ImpediMed Ltd, Brisbane, Australia).

SECONDARY OUTCOMES:
Interleukin 6 | Change from baseline to measurements taken daily for 7 days
  5mls blood from arterial catheter, centrifuged at 1,500 for 10 minutes at 4 degrees C. The supernaturant will be collected and stored at -80 degrees C. The marker will be analyzed by an enzyme-linked immuno-assay.
Tumour necrosis factor alpha (TNF-alpha) | Change from baseline to measurements taken daily for 7 days
  5mls blood from arterial catheter, centrifuged at 1,500 for 10 minutes at 4 degrees C. The supernaturant will be collected and stored at -80 degrees C. The marker will be analyzed by an enzyme-linked immuno-assay.
Interleukin 10 | Change from baseline to measurements taken daily for 7 days
  5mls blood from arterial catheter, centrifuged at 1,500 for 10 minutes at 4 degrees C. The supernaturant will be collected and stored at -80 degrees C. The marker will be analyzed by an enzyme-linked immuno-assay.
Vital signs - observation only | Fifteen minutes pre and post every exercise session recorded every 10 seconds
  Recording of vital signs ie heart rate, ECG, blood pressure, oxygen saturation from the IntelliVue bedside monitor MP70 (Phillips)

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Brisbane & Womens Hospital, Brisbane, Queensland, Australia